CLINICAL TRIAL: NCT00696566
Title: Study of the Potentiation of the Effects of Clopidogrel by Rifampicin in Healthy Volunteers
Brief Title: Healthy Volunteer Study of Clopidogrel and Rifampicin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: British Heart Foundation (Other); University of Sheffield (Other)
Responsible Party: Dr Robert Storey / Senior Lecturer & Honorary Consultant in Cardiology, University of Sheffield
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STH14468; BHF Grant: PG/05/095
Record Dates: First submitted 2008-06-04; First posted 2008-06-12 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Coronary Artery Disease
Keywords: Thrombosis; Platelet aggregation inhibitor; Blood platelets; P2 receptor; Cytochrome P450
MeSH Terms: conditions — Coronary Artery Disease; Thrombosis | interventions — Clopidogrel; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): All subjects will receive Clopidogrel and Rifampicin.
  Interventions: Drug: Clopidogrel and Rifampicin

INTERVENTIONS:
Drug: Clopidogrel and Rifampicin — Clopidogrel: loading dose of 600 mg, then 75 mg o.d. for up to 28 days
  Rifampicin: 300 mg b.d. for up to 28 days
  Other Names: Clopidorel = Plavix; Rifampicin = Rifadin

SUMMARY:
The principal research question is: Can platelet P2Y12 receptor blockade by the antithrombotic drug clopidogrel be significantly enhanced by coadministration of the antibiotic rifampicin?

Clopidogrel is an antithrombotic drug in clinical use that reduces the risk of heart attack and coronary stent thrombosis. However some patients respond poorly to clopidogrel, at least partly because they fail to convert it effectively to its active form, and consequently are at higher risk of arterial thrombosis. Preliminary evidence indicates that the antibiotic rifampicin enhances the effectiveness of clopidogrel by increasing its conversion to its active form by the liver. We wish to study further the extent of rifampicin's effect on clopidogrel to see whether this might be useful in clinical practice.

DETAILED DESCRIPTION:
Clopidogrel is an antithrombotic drug that is licensed for the treatment and prevention of arterial thrombosis, such as in people admitted to hospital with heart attacks. However, some people fail to achieve a substantial antithrombotic effect from the drug and one important reason for this is that their livers do not convert clopidogrel to its active form effectively. Current evidence suggests that these people are less protected by clopidogrel and have a higher risk of arterial thrombosis than those who respond well to clopidogrel. Rifampicin is an antibiotic that increases the activity of liver enzymes that convert clopidogrel to its active form and preliminary evidence indicates that it increases the effectiveness of clopidogrel. This raises the possibility that rifampicin might be used with clopidogrel to increase its clinical effectiveness. We wish to study this interaction further.

12 healthy volunteers will be recruited for this study after giving informed consent. Following Screening, the study will run over 28 days. Lab safety (clinical chemistry, haematology and urinalysis) will be undertaken on days 7, 22 and 28 in addition to screening. During the first visit, an intravenous cannula will be inserted into a forearm vein. Subjects will perform an erythromycin breath test. Subsequently, venous blood will be obtained via the intravenous cannula and platelet function studies will be performed and a plasma sample will be stored for baseline metabolite analysis. Subsequently the subjects will be administered a 600 mg loading dose of clopidogrel (Plavix, Sanofi Pharma Bristol-Myers Squibb) and further blood samples will be taken over 4 hours for clopidogrel metabolite analysis and platelet function studies. Subjects will then take clopidogrel 75 mg daily for a further 6 days and, 4 hours after the last dose, a further blood sample will be taken using venepuncture for platelet function studies and a plasma sample. After a washout period of 7 days, subjects will then start rifampicin 300 mg twice daily for 14 days (Rifadin, Aventis Pharma). On the 8th day of taking rifampicin, a further intravenous cannula will be inserted, the erythromycin breath test will be repeated, as above, and the same regimen of clopidogrel administration and blood testing will be repeated, this time with co-administration of rifampicin.

The data obtained will allow the following assessments: (i) comparison of the early effects of a 600 mg clopidogrel loading dose and late effects of clopidogrel after 7 days on platelet aggregation and receptor blockade; (ii) assessment of the effects of rifampicin on clopidogrel's action on platelet aggregation and receptor blockade following a loading dose and after prolonged administration of clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, or female subjects not of childbearing potential (either surgically sterile or post menopausal).
* Age between 18 and 65 years inclusive.
* Non smokers.
* Body mass index (BMI) between 18 and 28 kg/m2 inclusive, with a body weight between 60 - 100 kg.
* Subjects are to be in good health as determined by a medical history, physical examination including vital signs, and clinical laboratory test results including liver function and full blood count.
* Subjects have given their signed informed consent before any trial-related activity.

Exclusion Criteria:

* In the opinion of the investigator, subjects with, or a history of, cancer, diabetes or clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, haematological, dermatological, neurological, psychiatric or other major disorders.
* Subjects with a history of significant multiple drug allergies or with a known allergy to the study drugs or any medicine chemically related to the trial product.
* Subjects who have a clinically significant allergic disease (including hay fever).
* Subjects who have had a clinically significant illness within 4 weeks of dosing.
* Subjects taking regular medication including NSAID's, antibiotics, aspirin or anticoagulant therapy.
* Any clinically significant abnormal laboratory test results at screening.
* Subjects who have a supine blood pressure at screening, after resting for 5 min higher than 150/90 mmHg or lower than 100/50 mmHg.
* Subjects who have a supine heart rate at screening, after resting for 5 minutes outside the range of 40 - 90 beats/min.
* Subjects who have received any prescribed systemic or topical medication within two weeks prior to screening (although occasional use of paracetamol is permitted at the discretion of the investigator).
* Subjects who have received an investigational medicinal product within the previous four months (new chemical entity) or three months (licensed product) or subjects who have received a vaccine within three months preceding the start of dosing.
* Subjects who have donated any blood or plasma in the past month or in excess of 500 ml within twelve weeks preceding screening.
* Subjects who have a history of alcohol or drug abuse (consume greater than 28 units per week [one unit of alcohol equals 250 ml of beer or lager or one glass of wine or 20 ml of spirits]).
* Subjects with mental incapacity or language barriers which preclude adequate understanding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Can platelet P2Y12 receptor blockade by the antithrombotic drug clopidogrel be significantly enhanced by coadministration of the antibiotic rifampicin? | All year

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Storey, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Clinical Research Facility, Royal Hallamshire Hospital, Sheffield, S. Yorkshire, United Kingdom